CLINICAL TRIAL: NCT05390671
Title: Retrospective Analysis of the Use of CAR-T Cell Therapy in Patients With Hematological Malignancies in Spain
Brief Title: CAR-T Cell Therapy in Patients With Hematological Malignancies
Status: Completed | Type: Observational
Sponsor: Grupo Espanol de trasplantes hematopoyeticos y terapia celular (Other)
Responsible Party: Sponsor
Other Study IDs: GETH-CART-2020-01
Record Dates: First submitted 2022-04-27; First posted 2022-05-25 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: CART Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The prognosis of relapsed or refractory lymphoblastic leukaemia (ALL) and diffuse large B-cell lymphoma (DLBCL) is poor with conventional treatment with complete response rates around 25-30% with a median progression-free survival (PFS) of around 2 months and 7 months, respectively, despite the use of allogeneic and autologous haematopoietic stem cell transplantation. The recent introduction of CAR-T (Chimeric Antigen Receptor T-cells) therapy as a therapeutic option has been a breakthrough in the management of these entities.

DETAILED DESCRIPTION:
Information on baseline patient characteristics, haematological disease, comorbidities and CAR-T therapy procedure (lymphodepletion schedule, infused product) will be collected. Early post-infusion toxicity and recurrence data will be collected. The grading of adverse effects will follow the EBMT and ASTCT guidelines. Finally, data will be collected to analyse survival and, in case of death, cause of death).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients >18 y/o
* Patients receiving CAR-T cell therapy in Spain, since 2018.

Exclusion Criteria: T

* Patients receiving CART therapy as part of a clinical trial.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult patients >18, with hematologic malignancies (lymphoma, leukemia, myeloma) in which the use of CAR-T therapy is approved, undergoing CAR-T therapy in Spain.
Sampling Method: Probability Sample
Enrollment: 260 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Progression free survival | 6 month
  Patients who relapse or progress at 6 month after CART infussion.
Progression free survival | 12 month
  Patients who relapse or progress at 12 month after CART infussion.
Progression free survival | 24 month
  Patients who relapse or progress at 24 month after CART infussion.

SECONDARY OUTCOMES:
Overall survival | 6 month,12 month and 24 month
High relevance toxicity rates | During the firs month
  Rate of grade 3 or more of CRS and neurotoxicity
Progression free survival | 6 month,12 month and 24 month
  Patients who relapse or progress at 6, 12, 24 months from apheresis

CONTACTS AND LOCATIONS:
Locations (1):
- Angel Cedillo, Madrid, Spain